CLINICAL TRIAL: NCT07177456
Title: Study on the Safety and Efficacy of Umbilical Cord Blood Mononuclear Cells in the Treatment of Radiation-induced Lung Injury
Brief Title: Study on Safety and Efficacy of UCB-MNCs for Radiation-induced Lung Injury
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Zhu, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025&UCB-MNCs&RILI
Record Dates: First submitted 2025-09-09; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Radiation-induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCB-MNCs (Experimental): UCB-MNCs are obtained from umbilical cord blood by density gradient centrifugation
  Interventions: Biological: UCB-MNCs

INTERVENTIONS:
Biological: UCB-MNCs — UCB-MNCs were administered via intravenous infusion three times, once per week, with a dose of 3×10⁸ cells per infusion.

SUMMARY:
This study aims to evaluate the safety and efficacy of the umbilical cord blood mononuclear cells (UCB-MNCs) therapy for radiation-induced lung injuryr (RILI) by observing factors related to the therapeutic effect and adverse reactions of UCB-MNCs in treating RILI .

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-75 years,with no restriction on gender;
2. History of chest radiotherapy;
3. Diagnosed with grade 2-3 radiation-induced lung injury according to CTCAE 4.0 classification criteria in "Diagnosis and Treatment of Radiation-induced Lung Injury";
4. Inadequate response to conventional treatment for two weeks, with no relief or progressive worsening of symptoms;
5. Well-controlled tumor for ≥3 months;
6. No significant liver or kidney dysfunction: ALT, AST ≤ 3 times the upper limit of normal, serum Cr and BUN ≤ 2 times the upper limit of normal;
7. Expected survival ≥ 3 months;
8. Informed consent signed voluntarily by the patient;
9. Willing and able to receive treatment and follow-up as required by the protocol, and able to comply with basic treatment as directed by the physician.

Exclusion Criteria:

1. Severe cardiac insufficiency (such as NYHA class III or IV), uncontrolled hypertension (systolic blood pressure ≥160mmHg or diastolic blood pressure ≥110mmHg);
2. Positive for hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or syphilis;
3. ECOG score ≥2;
4. Currently participating in or participated in other clinical trials within 4 weeks;
5. History of allergies or known allergy to the study preparation;
6. Patients with psychiatric disorders who cannot cooperate with treatment; (7) Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Chest Enhanced CT Scan report | Baseline and at 1、3、6 and 12 months after the last treatment.
  Evaluate changes in lung damage ，and calculate the change in total lesion volume as a percentage of total lung volume.

SECONDARY OUTCOMES:
Modified Medical Research Council Dyspnea Scale (mMRC Score) | Baseline and at 1、3 、6 and 12 months after the last treatment.
  mMRC Score is a subjective scale for assessing the severity of breathing difficulties,dyspnea is classified into five grades (0 to 4). The higher the grade, the more severe the symptoms and the more obvious the limitation of movement.
6-minute walking distance test（6MWT） | Baseline and at 1、3 、6 and 12 months after the last treatment.
  The 6-minute walking distance (6MWD) is a method for assessing a patient's cardiopulmonary function and exercise endurance by measuring the maximum distance they can walk as fast as possible within 6 minutes.
Change from baseline in forced expiratory volume in 1st second (FEV1) | We measured FEV1 at baseline and at 1、3 、6 months and 12 months after the last treatment.
  FEV1 is the maximal volume of air that can be expired in 1st second of forced vital capacity maneuver using spirometry.
  We measured FEV1 at baseline and at 1、3 、6 months and 12 months after the last treatment.
Change from baseline in forced vital capacity (FVC) | We measured FVC at baseline and at 1、3 、6 months and 12 months after the last treatment.
  Forced vital capacity (FVC) is the maximal volume of air that can be expired while patient performs forced expiration as fast and as deep as possible using spirometry.
  We measured FEV1 at baseline and at 1、3 、6 months and 12 months after the last treatment.
Change from baseline in FEV1/FVC ratio | We measuredFEV1/ FVC at baseline and at 1、3 、6 months and 12 months after the last treatment.
  FEV1/FVC is used to differentiate obstructive from restrictive patterns by spirometry.
  We measuredFEV1/ FVC at baseline and at 1、3 、6 months and 12 months after the last treatment.
Change from baseline in lung Carbon Monoxide Diffusion Capacity (DLCO) | We measured DLCO at baseline and at 1、3 、6 months and 12 months after the last treatment.
  DLCO will be measured using the single breath-hold method with a Quark PFT gas analyzer, following ATS/ERS standards. Each test involves inhalation of a gas mixture (0.3% CO, 0.3% CH4, and dry air), breath-holding for 10±2 seconds, and exhalation.
  We measured DLCO at baseline and at 1、3 、6 months and 12 months after the last treatment.
Arterial blood gas parameter like pH value | We measured pH value at baseline and at 1、3 、6 months and 12 months after the last treatment.
  Compare pH value at baseline and at 1、3 、6 months and 12 months after the last treatment.
Arterial blood gas parameter like partial pressure of oxygen (PO2) | We measured PO2 at baseline and at 1、3 、6 months and 12 months after the last treatment.
  Compare the partial pressure of oxygen (PO2) at baseline and at 1、3 、6 months and 12 months after the last treatment.
Arterial blood gas parameter like oxygen saturation (SO2) | We measured SO2 at baseline and at 1、3 、6 months and 12 months after the last treatment.
  Compare the oxygen saturation (SO2) at baseline and at 1、3 、6 months and 12 months after the last treatment.
Arterial blood gas parameter like partial pressure of carbon dioxide (PCO2) | We measured PCO2 at baseline and at 1、3 、6 months and 12 months after the last treatment.
  Compare the partial pressure of carbon dioxide (PCO2) at baseline and at 1、3 、6 months and 12 months after the last treatment.

IPD SHARING:
Plan to Share IPD: No